CLINICAL TRIAL: NCT03934697
Title: In-Vivo Treatment for Imaginal Exposure Therapy
Brief Title: Imaginal Exposure II Study: In-Vivo
Acronym: In-vivo IE II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Cheri Levinson, Asst Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#:16.1003
Record Dates: First submitted 2018-10-16; First posted 2019-05-02 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Eating Disorder; Anorexia Nervosa; Bulimia Nervosa; Exposure
Keywords: Eating Disorder; Anorexia Nervosa; Bulimia Nervosa; Imaginal Exposure Therapy
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa | interventions — Implosive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaginal Exposure Session (Experimental): All participants will complete the same arm, which is ten sessions of imaginal exposure across a ten week time period. Each session is separated by 1 week.
  Interventions: Behavioral: imaginal exposure therapy

INTERVENTIONS:
Behavioral: imaginal exposure therapy — All participants will complete the same arm, which is ten sessions of imaginal exposure across a ten week time period. Each session is separated by 1 week.
  Other Names: Exposure Therapy

SUMMARY:
The purpose of this study is to test if imaginal exposure therapy can decrease symptoms of eating disorders and anxiety.

DETAILED DESCRIPTION:
An initial meeting consisting of a screening, questionnaires, and a brief psychoeducation on imaginal exposure therapy, followed by 8-10 sessions with a licensed psychologist (the PI) or a clinical psychology graduate student who is supervised and trained by the PI. In Session 1, patients will create a script with the therapist on an eating disorder fear. In sessions 2-10 the therapist and patient will then imagine this eating disorder related fear based on the script. Each session will be modified to focus on "hot spots" or the most feared aspect of the script. Sessions will be audiotaped and videotaped and participants will be asked to listen to the sessions nightly for homework. Sessions will be weekly or twice per week for 8-10 weeks after the initial screening session.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age (no age limit)
* Must currently meet criteria for anorexia, sub-clinical anorexia, bulimia, or sub-clinical bulimia (using the eating disorder diagnostic scale), OR have met criteria for one of these eating disorders in the last year, OR endorse significant eating disorder fears
* Must have at least one significant eating disorder related fear.

Exclusion Criteria:

* Under 18 years of age
* Individuals who have binge eating disorder or an unspecified eating disorder, OR who do not meet eating disorder related criteria
* Individuals who meet criteria for mania, psychosis, or suicidal ideation
* Participants who are not able to secure transportation to complete therapy sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-12-13 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
EDEQ (Eating Disorder Examination Questionnaire) at 1-10 Weeks and at 1 year | 1 year and 10 weeks
  The EDE-Q is a 41-item self-report questionnaire version of the Eating Disorder Examination, which is a semi-structured interview designed to assess eating disorders symptom frequency and severity over the past 28 days. The EDE-Q uses a 7-point forced-choice rating scheme (No days; 1-5 days; 6-12 days; 13-15 days; 16-22 days; 23-27 days; Everyday). The EDE-Q has four subscales with the question stem "How many days out of the past 28 days...": Restraint (e.g. Have you been consciously trying to restrict the amount of food you eat to influence your shape or weight?), Eating Concern (e.g. Have you had a definite fear that you might not be able to either resist eating or stop eating?), Weight Concern (e.g. Has your weight influenced how you think about (judge) yourself as a person?), and Shape Concern (e.g. How dissatisfied have you felt about your shape?).
SUDS (Subjective Units of Distress Scale) at 1-10 Weeks and at 1 year | 1 year and 10 weeks
  The SUDS scale is a self-report behavioral measure used during exposure treatment and behavioral assessment to measure anxiety. The SUDS scale has been shown to be a valid and reliable measure of state anxiety. SUDS ratings can range from 0 (completely calm) to 100 (highest anxiety). Other reference points used in this study include 25 (noticeable, but not bothersome anxiety), 50 (bothersome anxiety), and 75 (very bothersome anxiety). Subjective anxiety was assessed both in terms of categorical response and overall change. Categorical response was defined as a drop of at least five points in average SUDS across the exposure across visits.
Body Mass Index (BMI) at 1-10 Weeks and at 1 year | 1 year and 10 weeks
  Participants will be weighed at 1-10 Weeks and at 1 year and BMI will be calculated in order to see if the BMI of an individual has changed over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Eating Anxiety Treatment Laboratory and Clinic, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levinson CA, Rapp J, Riley EN. Addressing the fear of fat: extending imaginal exposure therapy for anxiety disorders to anorexia nervosa. Eat Weight Disord. 2014 Dec;19(4):521-4. doi: 10.1007/s40519-014-0115-6. Epub 2014 Apr 2. No abstract available. PMID 24691784
- [Background] Steinglass JE, Albano AM, Simpson HB, Wang Y, Zou J, Attia E, Walsh BT. Confronting fear using exposure and response prevention for anorexia nervosa: A randomized controlled pilot study. Int J Eat Disord. 2014 Mar;47(2):174-80. doi: 10.1002/eat.22214. Epub 2013 Nov 8. PMID 24488838
- [Background] Steinglass JE, Sysko R, Glasofer D, Albano AM, Simpson HB, Walsh BT. Rationale for the application of exposure and response prevention to the treatment of anorexia nervosa. Int J Eat Disord. 2011 Mar;44(2):134-41. doi: 10.1002/eat.20784. PMID 20127936